CLINICAL TRIAL: NCT04797871
Title: Resistance Training Intervention on the Clinical Status in Patients With Post Discharge Symptoms After Covid-19: The "EXER-COVID Study"
Brief Title: Resistance Training and Clinical Status in Patients With Post Discharge Symptoms After Covid-19
Acronym: EXER-COVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Pública de Navarra (Other)
Collaborators: Fundacion Miguel Servet (Other); Complejo Hospitalario de Navarra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: PI_2020/140
Record Dates: First submitted 2021-03-08; First posted 2021-03-15 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-07

CONDITIONS: Covid19; SARS-CoV2; Fatigue Syndrome, Chronic; Stress, Psychological; Pain, Chronic
MeSH Terms: conditions — COVID-19; Fatigue Syndrome, Chronic; Stress, Psychological; Chronic Pain | interventions — Resistance Training; Standard of Care

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Single (Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): Resistance training
  Interventions: Behavioral: Resistance training
- Standard care (Active Comparator): Non-supervised ACSM exercise guidelines
  Interventions: Behavioral: Standard care

INTERVENTIONS:
Behavioral: Resistance training — Participants will complete a 2-days-a-week training routine: Resistance training (RT, 50-75% 1RM (one-repetition maximum), 4 sets, 8-12 repetitions, 4 exercises). The warn up include Light Intensity Continuous Training (8-10 min, 65-70% HRR). Progressions will be individualized and consistent with patient tolerance. Sessions will be supervised by Physiotherapists and Graduated in Sports Sciences.
  Arms: Exercise
Behavioral: Standard care — This group will be allocated to standard care and therefore no supervised exercise regimen according to scientific guidelines for general physical activity and return to sport provided by the ACSM guidelines for Chronic Obstructive Pulmonary Disease and Cardiovascular Disease.
  Arms: Standard care

SUMMARY:
COVID-19 survivors commonly exhibit a marked extra-respiratory complication affecting the cardiac (arrhythmias and myocardial injury), renal (acute kidney injury), gastrointestinal, nervous (neuropathy, encephalopathy), endocrine and musculoskeletal (weakness, pain, and fatigue) systems. In this context, several studies have found that resistance training intervention promotes important health-related benefits, including cardiac function, compared to aerobic exercise training. Other exercise adaptations include increased skeletal muscle metabolism function, yet physio/psychological adaptations are known to be limited in COVID-19 survivors. Hence, given that resistance training intervention is implemented in a manner that is tolerable to the individual patient, it may be a potential beneficiary "personalized" rehabilitation treatment for patients with COVID-19 syndrome ambulatory.

The "EXER-COVID Clinical Study" project aims at determining the role of personalized exercise intervention in the treatment of post-COVID-19 syndrome ambulatory patients.

DETAILED DESCRIPTION:
100 patients will be recruited and undergo baseline testing, including examination, immune systems, biochemistry markers, ECG, DXA, metabolic/respiratory function, VO2max, muscular fitness, lipidomic/inflammatory/oxidative markers and psychological outcomes.

After baseline testing, participants will be randomly allocated into one group receiving standard of care (control group) or a group performing personalized resistance training intervention two times a week over a period of 6 weeks. The randomization procedure involves a computer-generated block randomization schedule in a ratio of 1:1 stratified by an independent person. Following the 8-week intervention period (with a 1-week washout period), both groups will complete a series of follow-up tests (as baseline testing). A 12-week follow-up experimental day is also planned in order to evaluate physio/psychological changes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* SARS-CoV-2 diagnosed using real-time reverse transcriptase polymerase chain reaction (PCR) tests or positive for SARS-CoV-2 virus antigen >90 days before randomization.
* Still present a chronic symptomatic phase lasting >90 days since debut of symptoms.
* Have not been hospitalized.
* There is no evidence on clinical records of pneumonia or any other organ failure related to SARS-CoV-2.
* Capable and willing to provide an informed consent.

Exclusion Criteria:

* Pregnancy or breast-feeding.
* Present atrial fibrillation.
* Diagnosed with acute myocarditis.
* Health conditions that prevent participating in the exercise intervention
* Patients who cannot undergo VO2max (e.g. acute heart attack or unstable angina, aortic stenosis, acute endocarditis / pericarditis, uncontrolled high blood pressure, acute thromboembolism, severe heart failure, respiratory failure and uncontrolled acute decompensated diabetes mellitus or low blood sugar).
* Treatment with IL-6 receptor antagonists (tocilizumab, kevzara) within the last month due to drug interference with the cardiopulmonary exercise adaptations.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2022-09-18 (Actual); Study Completion 2022-09-18 (Actual)

PRIMARY OUTCOMES:
Changes in Cardiorespiratory fitness | Baseline, 6 Weeks and 12 Weeks
  Measured with an incremental VO2 protocol on exercise bike by COSMED Quark CPET plus OMNIA (COSMED®, Rome, Italy)

SECONDARY OUTCOMES:
Changes in Post-COVID manifestations | Baseline, 6 Weeks and 12 Weeks
  Questionnaires that sought information about symptoms related to COVID-19 will be administrate. It is a dichotomous scale (Yes/No), that reflects symptoms, functional limitations, and clinical characteristics (i.e., nausea/vomiting, impaired visual acuity or blurry vision, anosmia, dizziness, depression, chills, weakness, musculoskeletal pain, palpitations/tachycardia, change of appetite, frustration, cognitive involvement, anxiety/irritability, dryness, impaired concentration, and headache)
Changes in Blood samples analysed for markers related to low grade inflammation | Baseline, 6 Weeks and 12 Weeks
  Including ENA-78, GCSF, GM-CSF, GRO, GRO-alpha, I-309, IL-1alpha, IL-1beta, IL-2, IL-3, IL-4, IL-5, IL-6, IL-7, IL-8, IL-10, IL-12 p40/p70, IL-13, IL-15, IFN-gamma, MCP-1, MCP-2, MCP-3, MCSF, MDC, MIG, MIP-1delta, RANTES, SCF, SDF-1, TARC, TGF-beta1, TNF-alpha, TNF-beta, EGF, IGF-I, Angiogenin, Oncostatin M, Thrombopoietin, VEGF-A, PDGF BB, Leptin in (arbitrary units).
Changes in pulse wave velocity | Baseline, 6 Weeks and 12 Weeks
  Measuring pulse wave velocity (m/seg) by VaSera VS 2000 (Fukuda Denshi, Japan)
Changes in cardio-ankle vascular index (CAVI) | Baseline, 6 Weeks and 12 Weeks
  Measuring Cardio-Ankle Vascular Index (%) by VaSera VS 2000 (Fukuda Denshi, Japan)
Changes in Energy expenditure | Baseline, 6 Weeks and 12 Weeks
  Measuring by COSMED Q-NRG+ plus OMNIA (COSMED®, Rome, Italy)
Changes in bone mineral density measured with DXA | Baseline, 6 Weeks and 12 Weeks
  Measuring in bone mineral density (g)
Changes in fat mass measured with DXA | Baseline, 6 Weeks and 12 Weeks
  Measuring in fat mass (%)
Changes in lean mass measured with DXA | Baseline, 6 Weeks and 12 Weeks
  Measuring in lean mass (kg)
Changes in Fat max oxidation rate | Baseline, 6 Weeks and 12 Weeks
  Measured with an incremental VO2 protocol on exercise bike by COSMED k-5 plus OMNIA (COSMED®, Rome, Italy)
Changes in Dynamic and isometric strength | Baseline, 6 Weeks and 12 Weeks
  Muscular fitness testing (legs, chest, arms, hip and grip)
Changes in Axial accelerometer-based physical activity monitors | Baseline, 6 Weeks and 12 Weeks
  Free-living physical activity is measured using axial accelerometer-based physical activity monitors (AX3; Axivity, Newcastle upon Tyne, UK)
Changes in blood samples analysed for markers related to oxidative stress | Baseline, 6 Weeks and 12 Weeks
  Including catalase, glutathione peroxidase, peroxidase, glutathione reductase in arbitrary units.
Changes in serum metabolic profiles | Baseline, 6 Weeks and 12 Weeks
  Utrahigh-performance liquid chromatography (UHPLC)-time of flight-MS based platforms analyzing methanol and chloroform/methanol serum extracts will be combined with the lipids measurement using an UHPLC-single quadrupole-MS based analysis in arbitrary units. Explained fraction of variance and the goodness of prediction will be calculated.
Changes in creatinine kinase | Baseline
  Creatinine kinase levels (units per liter)
Changes in total troponins levels (ng/mL) | Baseline
  Total troponins levels (ng/mL)
Changes in D-dimer | Baseline
  D-dimer (ng/mL)
Changes in thyroid function parameters | Baseline
  T3 and T4 levels (μg/dL)
Changes in liver function | Baseline
  ALT in (U/L), AST and GGT in (U/L)
Changes in renal function | Baseline
  Urea (mmol/L), sodium (mmol/L), potassium (mmol/L), chloride (mmol/L), calcium (mmol/L), inorganic phosphorus (mmol/L) and uric acid (mmol/L)
Changes in haematology parameters | Baseline
  White Blood Cells and Red Blood Cells (cell characterization)
Changes in cognitive status | Baseline, 6 Weeks and 12 Weeks
  Montreal Cognitive Assessment (MOCA) will be used as an indicator of cognitive status. Scores range between 0 and 30. A score of 26 or over is considered to be normal
Changes in visual attention and task switching | Baseline, 6 Weeks and 12 Weeks
  The Trail Making Test will be used as an indicator of visual scanning, graphomotor speed, and executive function. This test consists of two parts in which the subject is instructed to connect a set of 25 dots as quickly as possible while still maintaining accuracy
Changes in Quality of life | Baseline, 6 Weeks and 12 Weeks
  Two summary scores are reported from the EuroQOL EQ-5D instrument
Changes in psychological stress | Baseline, 6 Weeks and 12 Weeks
  The 1 Item Statistics Canada Stress Question (SCSQ) will be used. The SCSQ is a 1-item question with a possible scoring of 0 to 10, with higher scores indicating more stress.
Changes in physical health symptomology | Baseline, 6 Weeks and 12 Weeks
  A Physical Health item will be used in the baseline. The scoring range is 0-13, with higher numbers indicating experiencing more negative physical health symptoms.
Changes in psychological distress | Baseline, 6 Weeks and 12 Weeks
  The 10 Item Kessler Psychological Distress Scale will be used. Scores range from 10-50, with higher scores indicating more symptoms or more frequent experience of those symptoms.
Changes in depressive symptomology | Baseline, 6 Weeks and 12 Weeks
  The 10 Item Center for Epidemiologic Studies Depression Scale (CES-D) will be used in the baseline survey, and will be in each weekly survey to track changes in the CES-D over the study period. The possible range in scores is 0 to 30 depending on number of symptoms, with those symptoms weighted by frequency experienced in a week. Higher scores indicating more or more frequent symptoms.
Changes in life satisfaction | Baseline, 6 Weeks and 12 Weeks
  A Life Satisfaction item, consisting of three questions, will be used (scored 0-10). Higher scores indicate "the best possible life overall". In addition, 2-follow-up questions asking individuals to rate their physical and mental/emotional health on a five point scale from poor to excellent. Higher scores overall indicate more satisfaction with life.
Changes in resilience | Baseline, 6 Weeks and 12 Weeks
  The Brief Resilience Scale will be used (scores from 1-5). Higher scores indicate the individual perceives they have a better ability to 'bounce back' and recover from stressful events and/or situations.
Change in pain score using numeric 0-10 rating scale | Baseline, 6 Weeks and 12 Weeks
  The numeric rating scale is 0-10 where 0 is no pain, 5 is moderate pain and 10 is the worst pain
Tracking the amount of exercise variety participants feel they engage in | Baseline, 6 Weeks and 12 Weeks
  Using the Perceived Variety in Exercise questionnaire. There are 5 items asking about exercise variety, scored 1 (false) to 6 (true), with a possible score of 5-30; higher scores indicate greater perceived variety.
Changes in physical activity levels | Baseline, 6 Weeks and 12 Weeks
  Metabolic Equivalents (METs) throughout a week, including activity for work, during transport and leisure time, using the self-reported general physical activity questionnaire (GPAQ).
Including Changes in mononuclear cells of peripheral blood (sub-sample 40 participants) | Baseline, 6 Weeks and 12 Weeks
  CD4, CD8, PD1, CD62L, LKRG1, CD28, CD57, CD163, CD119, CD56, CD116, CD66b, CD11b, and CD14 by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Mikel Izquierdo, Ph.D, Study Chair — Universidad Publica de Navarra
Locations (1):
- Robinson Ramírez-Vélez, Ph.D, Pamplona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ramirez-Velez R, Oteiza J, de Tejerina JMCF, Garcia-Alonso N, Legarra-Gorgonon G, Oscoz-Ochandorena S, Arasanz H, Garcia-Alonso Y, Correa-Rodriguez M, Izquierdo M. Resistance training and clinical status in patients with postdischarge symptoms after COVID-19: protocol for a randomized controlled crossover trial "The EXER-COVID Crossover Study". Trials. 2022 Aug 9;23(1):643. doi: 10.1186/s13063-022-06608-y. PMID 35945634